CLINICAL TRIAL: NCT05661383
Title: Combining Hedonic Olfactory and BRAin Stimulations in Treatment-resistant Depression
Brief Title: Olfactory and Brain Stimulations in Treatment-resistant Depression
Acronym: COBRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-A01967-36
Record Dates: First submitted 2022-11-23; First posted 2022-12-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Treatment-resistant Depression
Keywords: Depression; brain stimulation; anhedonia; odor
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Anhedonia

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, randomized, double-blind, parallel-group controlled trial with two arms
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be block randomized (1:1) to receive either iTBS active combined with an olfactory stimulation or TBS active alone. Computer generated random numbers will be used to generate the allocation sequence. The allocation sequence will be handled by an independent person from the Administrative Department of the Hospital and will be unavailable to those who enroll and assign patients. Patients will be blind to their treatment assignment. Moreover, the medical doctors who will administer the clinical scales and the researchers that will analyze the data will be blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTBS active combined with an olfactory stimulation (Experimental): Non-invasive brain stimulation protocol (intermittent theta burst protocol (iTBS)) combined with pleasant odors delivered during the iTBS procol.
  Interventions: Device: Non-invasive brain stimulation protocol (intermittent theta burst protocol (iTBS)) combined with pleasant odors delivered during the iTBS procol.
- iTBS active alone (Active Comparator): Non-invasive brain stimulation protocol (intermittent theta burst protocol (iTBS)) delivered alone.
  Interventions: Device: Non-invasive brain stimulation protocol (intermittent theta burst protocol (iTBS)) delivered alone.

INTERVENTIONS:
Device: Non-invasive brain stimulation protocol (intermittent theta burst protocol (iTBS)) combined with pleasant odors delivered during the iTBS procol. — Device: MagPro X100 (MagVenture, Mag2Health, France) iTBS protocol targeting the left dorsolateral prefrontal cortex: 50 consecutive sessions allocated on 10 days (i.e., 5 sessions per working day, 1 hour apart, for 2 weeks).
  One iTBS session: burst of 3 pulses at 50 Hz repeated at 200 ms intervals for 2 s (i.e., at 5 Hz) at an intensity of 90% of rMT. A 2 s train of iTBS will be repeated every 10 s for a total of 1800 pulses per session.
  Pleasant odorants will be delivered using passive diffusers placed in the room dedicated to the iTBS protocol, during the all-treatment duration. During the inclusion phase, 10 odors known to be pleasant will be presented to the subject. The 3 best rated by the subject will be chosen for olfactory stimulations. During the iTBS session, a randomly selected odor from the 3 will be presented at the same time as the iTBS treatment.
  Arms: iTBS active combined with an olfactory stimulation
Device: Non-invasive brain stimulation protocol (intermittent theta burst protocol (iTBS)) delivered alone. — Device: MagPro X100 (MagVenture, Mag2Health, France) iTBS protocol targeting the left dorsolateral prefrontal cortex: 50 consecutive sessions allocated on 10 days (i.e., 5 sessions per working day, 1 hour apart, for 2 weeks).
  One iTBS session: burst of 3 pulses at 50 Hz repeated at 200 ms intervals for 2 s (i.e., at 5 Hz) at an intensity of 90% of rMT. A 2 s train of iTBS will be repeated every 10 s for a total of 1800 pulses per session.
  Arms: iTBS active alone

SUMMARY:
This is a prospective, randomized, double-blind, parallel-group controlled trial. The aim of this research project is to compare the clinical benefits achieved in patients with major depressive disorder (MDD) following two types of intervention: iTBS active alone or iTBS active combined with olfactory stimulations.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is the most widespread psychiatric disorder, affecting 5% of adults according to the World Health Organization. Anhedonia, defined as the loss of the ability to experience pleasure, is one of the key symptoms of depression, possibly due to a dysfunction of the reward system. Intermittent theta-burst stimulation (iTBS) targeting the dorsolateral prefrontal cortex (DLPFC) has been demonstrated as an emerging treatment option for treatment-resistant depression. One explanation is that iTBS could work through modulating the reward system (increasing dopamine release). One way to improve the therapeutic benefits of non-invasive brain stimulation is to combine it with other therapeutic strategies. Interestingly, olfactory training -daily short-term exposure to pleasant odors- improves significantly depressive symptoms in MDD patients. Indeed, the olfactory system and the reward system are closely related through the olfactory tubercle, which is in the ventral striatum and directly connected to the ventral tegmental area.

The general aim of this research project is to test whether a combination of iTBS targeting the left DLPFC with an olfactory training can improve treatment outcome in MDD, compared to iTBS targeting the left DLPFC alone.

The investigators hypothesize that combining iTBS treatment on DLPFC with hedonic olfactory stimulation potentiates the effect of iTBS treatment administered alone on depressive symptoms, especially anhedonia (physical, social or olfactory). Moreover, the investigators also hypothesize that the superiority of the combined approach is underpinned by greater modulation of connectivity activity and strength between brain regions involved in dopaminergic transmission, compared with iTBS alone.

ELIGIBILITY:
Inclusion Criteria:

* had a primary diagnosis of single-episode or recurrent non-psychotic major depressive disorder according to Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria;
* scored 20 or over on the MADRS (Montgomery-Åsberg Depression Rating Scale) (Montgomery and Åsberg, 1979) and scored higher than 2 on the MADRS item 8 anhedonia factor score;
* a stable antidepressant medication for 4 weeks prior to inclusion; be able to speak and read French;
* sign a consent form before intervention.

Exclusion Criteria:

* a pre-existing condition that affects olfaction including congenital anosmia, upper respiratory tract infection, nasal and/or sinus disease, brain injury or nasal surgery; a neurological disease;
* other comorbid psychiatric disorders or substance abuse (except tobacco);
* contraindications to TMS (medical devices implanted or metallic foreign body in the head);
* pregnant or lactating mothers (controlled by urine pregnancy tests);
* measure of protection or guardianship of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-27 (Actual); Primary Completion 2027-01-27 (Estimated); Study Completion 2027-10-02 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS score before and after intervention to characterized the number of depressed patients who reach remission criteria (MADRS ≤ 10) in each group | 4 times : before the Intervention (J0), immediately following the end of the Intervention (J15), 1 (M1) and 3 months (M3) after the end of the Intervention.
  MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to intervention. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
  Remission is defined as a Montgomery and Asberg Depression Rating Scale (MADRS) score less than or equal to 10 at the end of 50 sessions of iTBS

SECONDARY OUTCOMES:
Group differences in Montgomery-Asberg Depression Rating Scale (MADRS) score changes | 4 times : Before the Intervention (J0), immediately following the end of the Intervention (J15), 1 (M1) and 3 months (M3) after the end of the Intervention.
  MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to intervention. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores indicating a more severe depression.
Group differences in Beck Depressive Inventory (BDI) score changes | 4 times : before the Intervention (J0), immediately following the end of the Intervention (J15), 1 (M1) and 3 months (M3) after the end of the Intervention.
  BDI is a 21-item validated instrument for the self-report of depressive symptoms, with individual item scores summed to yield a total possible BDI score that ranges from 0-63. Higher scores indicating a more severe depression
Group differences in European Test of Olfactory Capabilities (ETOC) score changes | 2 times : Before the Intervention (J0), immediately following the end of the Intervention (J15)
  The ETOC is an olfactory test based on standardized odorants. It consists in the presentation of 16 odors at supraliminal concentrations. For each trial, 4 tubes are presented to the patient, but only one contains the odor. The participant has to find which one contains it. Then, the patient has to identify the odor between 4 propositions. Both tests are rated on 16. Another test will be performed to assess olfactory hedonic judgment. It consists of the presentation of 10 odors known to be pleasant. Hedonicity of each odor will be rated on an analog scale from 1 to 9 (1 for "Not at all pleasant", 5 for "Neutral" and 9 for "Extremly pleasant").
Group differences in the Chapman Social Anhedonia Scale (SAS) | 4 times : before the Intervention (J0), immediately following the end of the Intervention (J15), 1 (M1) and 3 months (M3) after the end of the Intervention.
  The SAS is a 40-items 'true/false' self-report questionnaire designed to measure social anhedonia that refers to a marked preference for solitary activities. Scores can range from 0 to 40 with higher scores indicating less ability to experience pleasure from social and interpersonal experiences.
the Chapman Physical Anhedonia Scale (PAS) score changes | 4 times : before the Intervention (J0), immediately following the end of the Intervention (J15), 1 (M1) and 3 months (M3) after the end of the Intervention.
  The PAS is a 61-items 'true/false' self-report questionnaire designed to measure physical anhedonia that refers to the inability to experience physical pleasures related to food, touch, smells, sex, temperature, movements, sounds and physical sensations. Scores can range from 0 to 61 with higher scores indicating less ability to experience pleasure from pleasant physical stimuli.
Group differences in conditioned motor evoked potential (MEP) peak-to-peak amplitude changes | 2 times : before the Intervention (J0), immediately following the end of the Intervention (J15)
  Dual-site transcranial magnetic stimulation (TMS) can be used to probe effective connectivity between the left DLPFC and the left M1. Conditioned MEP amplitude evoked by dual-site TMS and measured with surface EMG is compared to MEP amplitude evoked by TMS applied over M1 alone.
Group differences in functional connectivity changes in the targeted brain network | 2 times : before the Intervention (J0), immediately following the end of the Intervention (J15)
  Resting state functional magnetic resonance imaging (fMRI) is used to probe functional connectivity changes in the targeted brain region and related network following non-invasive brain stimulation intervention.
Group differences in the Childhood Trauma Questionnaire (CTQ) score changes | 1 time : Before the Intervention (J0)
  The CTQ is a self-administered 28-item scale to measure abuse and neglect suffered in childhood on five subscales: emotional, physical / sexual abuse, and emotional / physical neglect. Each subscale scored on a 5-point Likert scale. The score for each subscale classifies the severity of the abuse and neglect as: "none to minimal," "low to moderate," "moderate to severe" and "severe to extreme".

CONTACTS AND LOCATIONS:
Overall Officials: BRUNELIN JEROME, PhD, Principal Investigator — hospital le vinatier
Locations (1):
- CH Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided
Describe the IPD sharing plan, including what IPD are to be shared with other researchers.

REFERENCES:
- [Derived] Imbert L, Neige C, Dumas M, Bensafi M, Mandairon N, Brunelin J. Combining pleasant Olfactory and BRAin stimulations in treatment-resistant depression (COBRA): study protocol for a randomized controlled trial. Front Psychol. 2024 Dec 17;15:1451096. doi: 10.3389/fpsyg.2024.1451096. eCollection 2024. PMID 39744036